CLINICAL TRIAL: NCT07363369
Title: An Exploratory Basket Study on The Application of Therapeutic mRNA Vaccine Targeting FAP in Advanced Malignant Solid Tumors
Brief Title: Exploratory Clinical Study of FAP mRNA Vaccine in Patients With Advanced Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Liu, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-2148
Record Dates: First submitted 2026-01-12; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Tumors
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FAP mRNA vaccine, Dose 1 (Experimental): FAP mRNA vaccine
  Interventions: Biological: FAP mRNA vaccine (dose 1) + immune checkpoint inhibitors
- FAP mRNA vaccine, Dose 2 (Experimental): FAP mRNA vaccine
  Interventions: Biological: FAP mRNA vaccine (dose 2) + immune checkpoint inhibitors
- FAP mRNA vaccine, Dose 3 (Experimental)
  Interventions: Biological: FAP mRNA vaccine (dose 3) + immune checkpoint inhibitors
- FAP mRNA vaccine, Dose 4 (Experimental)
  Interventions: Biological: FAP mRNA vaccine (dose 4) + immune checkpoint inhibitors

INTERVENTIONS:
Biological: FAP mRNA vaccine (dose 1) + immune checkpoint inhibitors — FAP mRNA vaccine (dose 1) in combination with immune checkpoint inhibitors treatment
  Arms: FAP mRNA vaccine, Dose 1
Biological: FAP mRNA vaccine (dose 2) + immune checkpoint inhibitors — FAP mRNA vaccine (dose 2) in combination with immune checkpoint inhibitors treatment
  Arms: FAP mRNA vaccine, Dose 2
Biological: FAP mRNA vaccine (dose 3) + immune checkpoint inhibitors — FAP mRNA vaccine (dose 3) in combination with immune checkpoint inhibitors treatment
  Arms: FAP mRNA vaccine, Dose 3
Biological: FAP mRNA vaccine (dose 4) + immune checkpoint inhibitors — FAP mRNA vaccine (dose 4) in combination with immune checkpoint inhibitors treatment
  Arms: FAP mRNA vaccine, Dose 4

SUMMARY:
Cancer-associated fibroblasts (CAFs), as core regulators within the tumor microenvironment, significantly impede the intratumoral penetration of therapeutic agents and suppress the effective infiltration and activation of immune cells by constructing elaborate physical and functional barriers. Fibroblast activation protein (FAP) is a highly specific therapeutic target for CAFs, owing to its nearly tumor-restricted expression profile. Therefore, developing therapeutic strategies that specifically target FAP to eliminate CAFs and subsequently remodel the tumor microenvironment may effectively disrupt the multi-dimensional defense system established by CAFs, thereby significantly enhancing the delivery efficiency of anti-tumor agents and improving responsiveness to immunotherapy.

This Phase I clinical trial aims to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary antitumor activity of FAP mRNA Vaccine combined with immune checkpoint inhibitors in patients with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients: aged ≥ 18 years old;
* 2. Patients with histopathologically confirmed advanced malignant solid tumors (such as patients with advanced lung cancer, advanced colorectal cancer, advanced pancreatic carcinoma, etc.);
* 3. Patients refractory or intolerant to standard clinical treatment regimens;
* 4. According to the RECIST 1.1 criteria, at least one measurable lesion is required;
* 5. Eastern Cooperative Oncology Group (ECOG) performance status score: 0 - 1;
* 6. Expected survival time ≥ 3 months;
* 7. Main organ functions are in good condition;
* 8. Participants must have no plans for pregnancy during the treatment period and agree to use effective contraception voluntarily throughout the study period and for four months after discontinuation of treatment;
* 9. Sign a written informed consent form;
* 10. Ability to communicate effectively with the research team and willingness to comply fully with all protocol-specified requirements.

Exclusion Criteria:

* 1. History of other malignancies, except for adequately treated and non-recurrent within 5 years prior to screening basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, or gastrointestinal mucosal carcinoma, which the investigator deems eligible for inclusion;
* 2. Known central nervous system (CNS) metastases that are untreated or not effectively controlled by prior therapy;
* 3. Patients with serious cavity effusion;
* 4. Patient has comorbid conditions associated with elevated FAP expression beyond solid tumors, including pulmonary fibrosis, liver fibrosis, renal fibrosis, and rheumatoid arthritis, etc.;
* 5. Patients with uncontrolled cardiac clinical symptoms or diseases, such as heart failure of NYHA class II or above, unstable angina pectoris, having had a myocardial infarction within six months, and having clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention;
* 6. A history of thrombotic events (arterial or venous) within 6 months prior to enrollment, such as deep vein thrombosis, and pulmonary embolism;
* 7. Any active autoimmune disease or history of autoimmune diseases, including but not limited to: neurologic diseases related to immunity, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barré syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue disorders, scleroderma, inflammatory bowel disease (including Crohn's disease and ulcerative colitis), autoimmune hepatitis, toxic epidermal necrolysis (TEN), or Stevens-Johnson syndrome (excluding type 1 diabetes mellitus controlled with stable-dose insulin);
* 8. According to the investigator's judgment, there are concomitant uncontrolled diseases that may seriously endanger patient safety or affect the patient's completion of the study;
* 9. A known history of interstitial pneumonia or highly suspected interstitial pneumonia; or patients with lung abnormalities that could interfere with the detection or management of suspected drug-related pulmonary toxicity during the study;
* 10. Known allergy to the investigational drug (including any excipients). A history of severe allergic reactions to any drugs, foods, or vaccines, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, localized allergic necrotic reactions (Arthus reaction), etc.;
* 11. The last anti-cancer treatment occurred less than 4 weeks before the first vaccination; patients with unresolved treatment-related adverse effects (except hair loss) from previous anti-cancer treatments;
* 12. Patients who have previously received treatment with immune checkpoint inhibitors and experienced immune-related adverse events graded ≥3 according to the NCI CTCAE criteria;
* 13. Systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent doses of other glucocorticoids) or other immunosuppressive agents within 14 days before the first dose of the vaccine. However, the following situations are allowed: In the absence of active autoimmune disease, inhaled or local use of corticosteroids or adrenal hormone replacement with <=10 mg/day prednisone is allowed;
* 14. Received mRNA vaccines or lipid nanoparticles (LNP) or equivalent nanoparticle delivery drugs within 6 months prior to the first dose of the vaccine;
* 15. Previously received live attenuated vaccine/inactivated vaccine within 6 months;
* 16. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 17. Blood donation or significant blood loss (>450 mL) within 3 months prior to screening;
* 18. Major surgery within 4 weeks prior to screening (small surgeries such as catheter placement, biopsy required by the protocol, etc., are not exclusion criteria), or the surgical or traumatic effects have not been resolved within 14 days before enrollment;
* 19. A history of drug abuse or known medical, psychological, or social conditions, such as a history of alcoholism or drug abuse;
* 20. Human immunodeficiency virus (HIV) positive, or positive for syphilis antibodies; patients with active HBV infection, or HCV infection;
* 21. Patients with active tuberculosis (TB) or a history of active TB; or those requiring systemic treatment for severe acute or chronic infections
* 22. Pregnant or breastfeeding women;
* 23. Any other factors that the investigator believes may make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) and their incidence rates | During one year after initial treatment
Safety: Type, frequency, and severity of treatment-related adverse events as assessed by CTCAE V5.0 | During one year after initial treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | During one year after initial treatment
Disease control rate (DCR) | During one year after initial treatment
Progression-free survival (PFS) | During one year after initial treatment
Immunogenicity: Specific T cell levels targeting FAP antigen | During one year after initial treatment